CLINICAL TRIAL: NCT05522114
Title: Evaluation of Patient Specific Guide Accuracy for TMJ Superior Joint Space Injection.
Brief Title: Accuracy of Patient Specific Guide for TMJ Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, AbdElKader Ahmed Hyder Mohamed, Principal Investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSG-TMJ-acc.
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: TMD
Keywords: virtual planning; 3D printing; TMD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient specific guided injection (Experimental): Patients treated with HA injection in TMJ using PSG and the accuracy evaluated using MSCT.
  Interventions: Procedure: TMJ injection using patient specific guide

INTERVENTIONS:
Procedure: TMJ injection using patient specific guide — Prefabricated patient specific guide used to guide the needle into the superior joint space of TMJ while real time MSCT evaluate the accuracy of needle position. Sodium hyaloronate injected within the superior joint space.

SUMMARY:
This study is designed to evaluate the accuracy of planned needle position using patient specific guide during TMJ superior joint space injection.

DETAILED DESCRIPTION:
The actual position of the needle evaluated in comparison to the planned one using MSCT while the patient wearing the customized needle guide.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with intra-articular TMJ disorder according to Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD).
* Patients who would not respond to conservative treatment as the first line of treatment.

Exclusion Criteria:

* Lactating, pregnant or planning pregnancy women.
* Known hypersensitivity to hyaluronic acid or clear biocompatible photopolymer resin.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Angle of deviation | 1 month
  The angle (°) between the planned and actual needle measured.
Vertical displacement of needle tip | 1 month
  The vertical displacement of the actual needle tip in comparison to the planned one (mm).
Overall needle tip dislocation | 1 month
  The distance between the planned and actual needle tips (mm).

CONTACTS AND LOCATIONS:
Overall Officials: AbdElKader A Hyder, MSc, Principal Investigator — Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Al-Azhar University; Wael A ElMohandes, PhD, Study Director — Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Al-Azhar University; Bahaa El-Din A Tawfik, PhD, Study Director — Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Al-Azhar University
Locations (1):
- Faculty of Dentistry, Al-Azhar University., Cairo, Egypt